CLINICAL TRIAL: NCT06613490
Title: An Exploratory Clinical Study of the Safety and Efficacy of CD19 Chimeric Antigen Receptor NK Cells for the Treatment of Refractory Antisynthetase Antibody Syndrome and Rheumatoid Arthritis
Brief Title: An Exploratory Clinical Study of CD19 CAR NK Cells for the Treatment of Refractory Antisynthetase Antibody Syndrome and Rheumatoid Arthritis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, Wenfeng Tan, Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-834
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Antisynthetase Syndrome; Rheumatoid Arthritis
MeSH Terms: conditions — Antisynthetase syndrome; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti CD19 CAR NK cells (Experimental)
  Interventions: Biological: anti CD19 CAR NK cells

INTERVENTIONS:
Biological: anti CD19 CAR NK cells — This study is a single-arm, open-label and single-center exploratory clinical study to evaluate the safety and effectiveness of anti CD19 CAR NK cells in patients with refractory antisynthetase antibody syndrome (ASyS) and rheumatoid arthritis (RA). All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by Anti-CD19 CAR NK cells infusion.

SUMMARY:
A single-center, open-label dose-escalation design to evaluate the safety and efficacy of 3 infusions of anti CD19 CAR NK cells (KN5501), as well as the expansion and persistence of KN5501 in patients with refractory antisynthetase antibody syndrome (ASyS) and rheumatoid arthritis (RA); To evaluate the ability of KN5501 to clear CD19-positive B cells in patients to determine the feasibility of KN5501 for the treatment of refractory ASyS and or RA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign the Informed Consent Form (ICF) , participate in this clinical study and be willing to follow and be able to complete all trial procedures.
2. Defined according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria, adult patients with RA diagnosed ≥3 months prior to screening;Moderately to severely active RA;Poor response, or loss of response, or intolerance to at least one conventional synthetic DMARD (csDMARD) or biologic DMARD (bDMARD) or targeted synthetic DMARD (tsDMARD).
3. Defined according to the 2020 ENMC-DM classification diagnostic criteria. Adult patients with ASyS diagnosed ≥3 months prior to screening; patients with moderately severe active ASyS.
4. Age: ≥ 18 years old and ≤ 70 years old, male or female.
5. Subjects with estimated survival > 12 weeks.
6. Serum creatinine clearance meets the relevant age/sex criteria, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN).
7. ECOG score 0 - 2.
8. The heart structure is essentially normal by echocardiography and Left ventricular ejection fraction (LVEF) ≥45%.
9. 2 weeks after the subject received the last dose treatment (hormonal, immunosuppressive or other experimental treatment).

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions.
2. Subjects with one of the following genetic syndromes: Fanconi syndrome, Kostmann syndrome, Shwachman syndrome or any of the known bone marrow failure syndromes.
3. Subjects with Active or uncontrolled infections requiring parenteral antimicrobials; evidence of severe active viral or bacterial infections or uncontrolled systemic fungal infections.
4. Subjects with grade III or IV heart failure (NYHA classification).
5. History of epilepsy or other central nervous system (CNS) diseases.
6. Subjects with history of malignancy except cured of carcinoma in situ of the skin or cervix, and patients with inactive tumors.
7. Subjects with pronounced bleeding tendencies, such as gastrointestinal bleeding, coagulation disorders, and hypersplenism.
8. The subject with unstable angina, symptomatic congestive heart failure or myocardial infarction within the last 6 months.
9. Females who are pregnant, lactating, or planning a pregnancy within six months.
10. Subjects who have received other clinical trial treatment within 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 52 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5501) for refractory antisynthetase antibody syndrome (ASyS) and rheumatoid arthritis (RA)
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 52 weeks after infusion
  To characterize the safety of CD19 CAR NK Cells (KN5501) for refractory antisynthetase antibody syndrome (ASyS) and rheumatoid arthritis (RA)

SECONDARY OUTCOMES:
The overall response rate (ORR) | 4, 12, 24, 36 and 52 months after infusion
  To characterize the efficacy of CD19 CAR NK Cell (KN5501) for refractory antisynthetase antibody syndrome (ASyS) and rheumatoid arthritis (RA)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No